CLINICAL TRIAL: NCT07101562
Title: Clinical Transformation of Bone Reconstruction With Autologous Bone Marrow Mesenchymal Stem Cells in Vitro to Repair Avascular Necrosis of Femur Head
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEBANFH-2023
Record Dates: First submitted 2025-06-25; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Avascular Necrosis of Femur Head
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tissue-engineered bone to repair Avascular Necrosis of Femur Head (Experimental): Tissue-engineered bone with autologous bone marrow mesenchymal stem cells to repair Avascular Necrosis of Femur Head
  Interventions: Device: Tissue-engineered bone

INTERVENTIONS:
Device: Tissue-engineered bone — Tissue-engineered bone with autologous bone marrow mesenchymal stem cells

SUMMARY:
The commercial decalcified bone scaffold combined with the patient's autologous bone marrow mesenchymal stem cells was used for in vitro culture to form tissue-engineered bone, and the effect of this tissue-engineered bone in early non-traumatic femoral head necrosis was explored.

DETAILED DESCRIPTION:
Avascular necrosis of the femoral head progresses rapidly, and most patients experience femoral head collapse within 1 to 4 years. Therefore, early intervention in the early stage of avascular necrosis of the femoral head is crucial for preserving the femoral head. Currently, core decompression is commonly used in clinical practice for early avascular necrosis of the femoral head. The principle is to drill holes and partially remove the necrotic lesions to reduce the pressure within the femoral head, increase blood supply, stimulate bone regeneration, thereby alleviating pain and delaying or reversing the progression of avascular necrosis of the femoral head. After the necrotic area of the femoral head is removed, bone grafting is often required to prevent complications such as femoral neck instability, femoral neck fractures, and femoral head collapse. There are many types of bone grafts, such as autologous bone, allogeneic bone, and artificial bone. However, autologous bone causes damage to the donor site and provides limited bone tissue; allogeneic bone has limited bone repair ability due to the lack of biological activity. Tissue engineering technology uses tissue engineering methods to transplant a composite of seed cells, growth factors, and scaffold materials to the bone defect site, providing good structural support and promoting bone tissue regeneration, thereby repairing the necrotic area of the bone and blood vessels. It has the advantages of no rejection reaction, unrestricted material acquisition, sufficient bone mass for cultivation, and easy survival, providing a new direction for the treatment of avascular necrosis of the femoral head. This study aims to evaluate the clinical effect of tissue-engineered bone in repairing early non-traumatic aseptic necrosis of the femoral head and provide a basis for the treatment of aseptic necrosis of the femoral head.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and voluntarily signing the informed consent form before the study;
2. Meets the diagnostic criteria in the "Clinical Diagnosis and Treatment Guidelines for Adult Femoral Head Necrosis in China (2020)";
3. Age range: 20 - 65 years old (inclusive of boundary values), gender not restricted;
4. Staged as ARCO II stage;
5. Non-traumatic femoral head necrosis;
6. Has received conservative treatment (such as physical therapy, blood-activating, analgesic drugs, etc.) for more than 2 weeks, and the target hip joint still shows persistent pain symptoms;
7. The subjects are usually able to move, not bedridden or in a wheelchair for a long time, and can walk more than 50 meters without the help of crutches or walking sticks;
8. During the trial period and within 90 days after the surgery, the subjects have no pregnancy plans and voluntarily take effective contraceptive measures.

Exclusion Criteria:

1. Based on the researcher's judgment, the subjects had a history of trauma and the injury affected the target hip joint;
2. In the six months prior to screening, there were obvious injuries involving the target hip joint;
3. The subject's femoral head necrosis was due to other diseases affecting the hip joint (such as rheumatoid arthritis, psoriatic arthritis, gouty arthritis, symptomatic cartilage calcification, bone necrosis, active infection), or according to the researcher's judgment, peripheral or central nervous system lesions that might affect the assessment of pain and function of the target hip joint (such as back pain, knee joint disease, intervertebral disc protrusion, sciatic nerve pain, fibromyalgia, diabetic neuropathy, etc.);
4. The femoral head of the target hip joint had obvious necrosis, collapse, joint fusion, etc.;
5. Those who had a history of hip joint replacement, arthroplasty, or other hip joint surgeries, or planned to undergo surgical treatment of any lower limb/hip joint during the study period;
6. The target hip joint had suppurative arthritis or a previous history;
7. The target hip joint had obvious joint effusion;
8. During the screening period, the target hip joint had active joint infection or skin ulceration, infection in the surgical area, or any significant chronic skin disease that might interfere with the surgical procedure;
9. The subject was treating the target hip joint, and within 30 days before screening, had used opioids or glucocorticoids for treatment; or was required to use opioids or glucocorticoids for long-term treatment during the study period;
10. Patients who had received any drug injection or surgical treatment in the hip joint (both sides or any one side) within 6 months before the treatment start;
11. Started using drugs such as cilostazol for promoting blood circulation and anticoagulation therapy 8 weeks before screening;
12. Note: If antihypertensive drugs or anticoagulant drugs such as cilostazol were used for treatment for ≥ 8 weeks before screening, they could be used at a stable dose during the study period;
13. The subject had a disease requiring systemic glucocorticoid treatment;
14. Abnormal liver and kidney function: At the time of screening, AST or ALT > 2 × upper limits of normal (ULN); or serum creatinine > 1.5 × ULN, or creatinine clearance rate ≤ 50 mL/min;
15. Note: For men, the creatinine clearance rate (mL/min) = [(140 - age) × weight (kg)] / [0.818 × Cr (μmol/L)]; for women, the creatinine clearance rate (mL/min) = male creatinine clearance rate (mL/min) × 0.85;
16. The subject had any type of active malignant tumor and was receiving systemic chemotherapy; or within 5 years before screening, was diagnosed with cancer (excluding squamous cell carcinoma or basal cell carcinoma of the skin);
17. According to the researcher's judgment, before enrollment, 12-lead electrocardiogram (ECG) showed clinically significant abnormalities; including QTc (QTcB) > 450 ms, or heart rate > 100 bpm, or QRS > 120 ms, or PR > 220 ms;
18. Basic cardiovascular diseases: Within 6 months before enrollment, had experienced the following cardiovascular events: myocardial infarction or coronary artery bypass surgery or traumatic coronary artery reperfusion surgery or stroke; unstable angina pectoris; variant angina pectoris; symptomatic congestive heart failure (New York Heart Association cardiac function grade III-IV or ejection fraction ≤ 35%);
19. Uncontrolled hypertension (defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg after standardized antihypertensive drug treatment);
20. Positive hepatitis B surface antigen, hepatitis C antibody, AIDS antibody, syphilis antibody tests;
21. Those who are known or suspected to be allergic to the active or inactive ingredients of the research drug;
22. Gastrointestinal underlying diseases: having a history of gastrointestinal bleeding or perforation after using non-steroidal anti-inflammatory drugs (NSAIDs); subjects with active gastrointestinal ulcer bleeding within 30 days before enrollment, or who have had recurrent ulcer bleeding in the past;
23. Allergic to the test drug or having a history of hypersensitivity reaction;
24. Subjects unable to avoid non-habitual physical activities (such as starting new weightlifting exercises);
25. Having a clear history of mental disorder, or having a history of abuse of psychotropic drugs or drug addiction;
26. Alcohol (defined as drinking more than 2 units per day/ more than 14 units per week, 1 unit being equivalent to 360ml of beer or 45ml of 40% alcohol content spirits or 150ml of wine) or drug abusers; or those with mental disorders;
27. Pregnant women, lactating women, and women of childbearing age who have not undergone sterilization surgery/are not in menopause/are unwilling to use medically approved effective contraceptive measures during the study period; men who have not undergone sterilization surgery/are unwilling to use medically approved effective contraceptive measures during the study period;
28. Those who have participated in any other clinical trials within 3 months before screening;
29. Other situations deemed unsuitable for participation in this trial by the investigator.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To verify the effectiveness of tissue-engineered bone in the treatment of early femoral head necrosis | 1 month, 2 months, 3 months, 6 months and one year after the operation
  The judgment is mainly based on the X-ray plain films and MRI results of the hip joint during the follow-up process: ① Improvement: New bone is generated in the necrotic bone tissue within the femoral head; ② Unchanged: There was no further collapse of the femoral head; ③ Deterioration: Femoral head collapses, osteoarthritis occurs in the femoral head, and total hip replacement arthroplasty (THA) is performed. If the imaging indicates improvement or no change, the imaging is successful; if it indicates deterioration, it is a failure.
To verify the effectiveness of tissue-engineered bone in the treatment of early femoral head necrosis | Before the operation, 1 month, 6 months and 1 year after the operation
  The degree of pain of the patients was evaluated by visual analogue scales (VAS) before the operation, 1 month, 6 months and 1 year after the operation respectively. The VAS pain score standard: A score of 0 to 10, from low to high, indicates an increase in the degree of pain. A score of 0 indicates no pain, and a score of 10 indicates severe and unbearable pain.
To verify the effectiveness of tissue-engineered bone in the treatment of early femoral head necrosis | Before the operation, 6 months after the operation and 1 year after the operation
  The hip joint function of the patients was evaluated by Harris score before the operation, 6 months after the operation and 1 year after the operation respectively. The total score of the Harris score is 100 points, including 44 points for the pain score, 51 points for the functional score (daily activities, walking gait, walking distance, degree of deformity), and 5 points for the range of motion of the hip joint (forward flexion, abduction, external rotation, adduction, internal rotation).

SECONDARY OUTCOMES:
Verify the safety of tissue-engineered bone | 1 month, 2 months, 3 months, 6 months and one year after the operation
  Number of participants with adverse events/serious adverse events, with abnormal laboratory tests results, abnormal vital signs, abnormal physical examination and abnormal electrocardiogram readings

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan, China